CLINICAL TRIAL: NCT02101177
Title: Evaluation of the National Treatment Program of Hepatitis C in Egypt, Using Data Coming From Two Treatment Centres.
Brief Title: Evaluation of the National Treatment Program of Hepatitis C in Egypt
Acronym: eNTC
Status: Withdrawn | Type: Observational
Why Stopped: Study objectives were considered as absolete regarding the arrival of new antiviral drugs in Egypt.
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut Pasteur (Industry); National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12291
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Hepatitis C
Keywords: Viral Hepatitis C; Genotype 4; SVR; Egyptian National Program
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — * Plasma
  * Serum
  * PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients under Dual therapy: - 1500 patients who started treatment between April 1st 2013 and March 31st 2014 and will be seen for their week 60 visit between July 1st 2014 and June 30th 2015 (Cohort A).
- Early Defaulters: - 1000 patients recruited between July 1st 2014 and estimated March 31st 2015, of which 200 are expected to be early defaulters and will be contacted by the study team (Cohort B).

SUMMARY:
The aim of the study is to analyse data coming from two treatment centres of the National Treatment Program Centres of hepatitis C in Egypt

DETAILED DESCRIPTION:
Analyse data coming from two centres of the National Treatment Program of hepatitis C in Egypt:

* 1500 patients who started treatment between April 1st 2013 and March 31st 2014 and will be seen for their week 60 visit between July 1st 2014 and June 30th 2015 (Cohort A).
* 1000 patients recruited between July 1st 2014 and estimated March 31st 2015, of which 200 are expected to be early defaulters and will be contacted by the study team (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years and > 60 years
* Positive HCV antibodies using a third generation test
* Detectable HCV RNA by PCR
* Liver biopsy showing chronic hepatitis with either a METAVIR score F1 with elevated liver enzymes or scores F2/F3
* Naïve to treatment with PEG-IFN and RBV
* HBs antigen negative
* Prothrombin time ≥60 %, normal bilirubin, alpha-foeto protein < 3*normal range of the laboratory, anti-nuclear antibodies<1/160
* Effective contraception during the treatment period; no breast-feeding
* Signed informed consent and willingness to participate in the study

Exclusion Criteria:

* Serious co-morbid conditions such as severe hypertension, heart failure, significant coronary heart disease, poorly controlled diabetes (HbA1C>8%) , chronic obstructive pulmonary disease
* Major uncontrolled depressive illness
* Solid transplant organ (renal, heart, or lung)
* Untreated thyroid disease
* History of previous anti-HCV therapy
* Body mass index (BMI) greater than 30 kg/m²
* Known human immunodeficiency virus (HIV) coinfection: although HIV testing will not be proposed or done, patients with known HIV coinfection will not be included in the trial
* hypersensitivity to one of the two drugs (PEG-IFN, RBV)
* pregnancy or unwilling to comply with adequate contraception
* breast-feeding
* neutropenia (<1500/mm3)
* anaemia (<11g/dL for women ; <12g/dL for men)
* thrombocytopenia (<100.000/mm3)
* elevated creatinin (>1.5mg/dL)
* concomitant liver disease other than hepatitis C (immuno-active chronic hepatitis B, autoimmune hepatitis, alcoholic liver disease, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson disease)
* liver biopsy showing severe steatosis (>66%) and steatohepatitis; decompensated cirrhosis (Child Pugh>A); hepatocellular carcinoma, METAVIR score F4.
* TSH>5 mU/L

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients included in the study will be those with prior approval from the Ministry of Health to begin the bi-therapy and attending two centres of the National Treatment Program.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Estimate "real life" Sustained Virological Response rate | 60 weeks after initiation of treatment
  Put in place mechanisms to ensure systematic reporting of HCV RNA testing at week 60 in the two project centres to obtain reliable estimates of response rates at this crucial time point.

SECONDARY OUTCOMES:
Compare the efficacy of Reiferon®, a biosimilar produced by a local company, Minapharm©, to that of other pegylated interferon of known efficacy (Pegasys®, Pegintron®) | 12 weeks, 24 weeks and 60 weeks after initiation of treatment
  Response rates at week 12, week 24 and week 60 will be compared across the three treatment regimens available in Egypt. Reiferon's efficacy will be assessed by comparison of:
  * Complete early virological response (cEVR): defined by undetectable HCV RNA at 12 weeks post initiation of dual therapy by PEG IFN + RBV
  * Early virological response (EVR): defined by at least a 2 log-reduction of HCV RNA or undetectable HCV-RNA at 12 weeks of combination therapy.
  * Sustained virological response (SVR): defined by HCV RNA below the detection limit based on quantitative PCR 12 weeks after stopping treatment (week 60)
  * Normalization of ALT: Proportion of patients who have ALT below the upper limit of normal (ULN) during the treatment and 12 weeks after the end of treatment.
  * Adverse events: Evaluation of Incidence of AE and SAE related to dual therapy.
Understand the determinants of not returning for follow-up among defaulting patients | 60 weeks after the initiation of dual-therapy
  Describe the timing of premature termination of treatment, and understand factors associated with it, throughout the 60 weeks of follow-up. Patients compliance in terms of regularity of injections intake will be described
Optimize selection criteria for patients to be enrolled in the National Treatment Program | 60 weeks after the initiation of dual therapy
  Explore various inclusion criteria combining fibrosis stage and serological markers of treatment response to optimize the selection of patients for the National Treatment Program
Estimate "real life" Response rate at the end of treatment | 48 weeks after initiation of treatment
  Put in place mechanisms to ensure systematic reporting of HCV RNA testing at week 48 in the two project centres to obtain reliable estimates of response rates at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wahid DOSS, MD, PhD, Principal Investigator — National Hepatology & Tropical Medicine Research Institute; Arnaud FONTANET, MD, PhD, Principal Investigator — Institut Pasteur
Locations (2):
- Egypt (2):
  - El Fahera El Fatemia, Cairo
  - NHTMRI, Cairo

REFERENCES:
- [Background] Breban R, Doss W, Esmat G, Elsayed M, Hellard M, Ayscue P, Albert M, Fontanet A, Mohamed MK. Towards realistic estimates of HCV incidence in Egypt. J Viral Hepat. 2013 Apr;20(4):294-6. doi: 10.1111/j.1365-2893.2012.01650.x. Epub 2012 Sep 13. PMID 23490375
- [Background] Guerra J, Garenne M, Mohamed MK, Fontanet A. HCV burden of infection in Egypt: results from a nationwide survey. J Viral Hepat. 2012 Aug;19(8):560-7. doi: 10.1111/j.1365-2893.2011.01576.x. Epub 2012 Feb 6. PMID 22762140
- [Background] El Makhzangy H, Esmat G, Said M, Elraziky M, Shouman S, Refai R, Rekacewicz C, Gad RR, Vignier N, Abdel-Hamid M, Zalata K, Bedossa P, Pol S, Fontanet A, Mohamed MK. Response to pegylated interferon alfa-2a and ribavirin in chronic hepatitis C genotype 4. J Med Virol. 2009 Sep;81(9):1576-83. doi: 10.1002/jmv.21570. PMID 19626613
- See also: Egyptian National Control Strategy For Viral Hepatitis (2008-2012) — http://www.hepnile.org/index.php/national-strategy-document